CLINICAL TRIAL: NCT01303263
Title: A Brief Intervention to Improve Cost-effective Resource Use Among Medicine Housestaff
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Partners Center of Expertise in Quality and Patient Safety (Unknown)
Responsible Party: David Bates, Brigham & Women's Hospital
Allocation: Randomized
Other Study IDs: 2009-P-001758/1; BWH
Record Dates: First submitted 2011-02-23; First posted 2011-02-24 (Estimated); Last update posted 2011-06-22 (Estimated); Status verified 2011-02

CONDITIONS: Graduate Medical Education; Cost-Effectiveness
Keywords: efficiency; cost-awareness; hospitals; graduate medical education
MeSH Terms: interventions — Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Group (Other): Residents Randomized to Receive Educational Intervention
  Interventions: Behavioral: Educational Intervention
- Control Group (No Intervention): Residents randomized not to receive a teaching intervention.

INTERVENTIONS:
Behavioral: Educational Intervention — 45-minute teaching session on healthcare costs, in which each resident reviewed an itemized hospital bill for a patient he/she had cared for, followed by an open-ended discussion about reducing unnecessary costs.
  Arms: Intervention Group

SUMMARY:
OBJECTIVE: To test a brief intervention designed to improve the cost-effectiveness of care provided by medicine housestaff for hospitalized patients.

HYPOTHESIS: A brief intervention in which medicine residents receive itemized bills for recent patients cared for by them, followed by a discussion on approaches to reducing unnecessary inpatient costs, can result in significant cost reductions without adversely affecting patient outcomes.

DETAILED DESCRIPTION:
We designed a brief educational intervention with two primary objectives: 1) to increase awareness among residents about how their decisions impact the costs of inpatient medical care; and 2) to improve the cost-effectiveness of care provided by residents without adversely affecting patient outcomes. We hypothesized that a brief intervention in which residents receive bills for patients they recently cared for, followed by a discussion on approaches to reducing unnecessary inpatient costs, would reduce costs without adversely affecting patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Internal Medicine Residents on Inpatient Rotations at Brigham & Women's Hospital

Exclusion Criteria:

* Having a team member who was in either the control group or intervention group in a prior round of this study.

Sex: All
Age Groups: Child, Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2009-09; Primary Completion 2010-12 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Total Cost | 2 weeks following educational intervention
  Total hospital cost per admission for 2 weeks following the educational intervention.
Lab Cost | 2 weeks following educational intervention
  Total lab cost per admission for 2 weeks following the educational intervention.
Pharmacy Cost | 2 weeks following educational intervention
  Total pharmacy cost per admission for 2 weeks following the educational intervention.
Radiology Cost | 2 weeks following educational intervention
  Total radiology cost per admission for 2 weeks following the educational intervention.

SECONDARY OUTCOMES:
length of stay | 2 weeks after educational intervention
admission to an intensive care unit (ICU) | 2 weeks after educational intervention
30-day readmission | within 30 days after end of study period
30-day mortality | within 30 days after end of study period

CONTACTS AND LOCATIONS:
Overall Officials: David Bates, MD, Principal Investigator — Brigham and Women's Hospital; Benjamin D Sommers, MD, PhD, Study Director — Brigham and Women's Hospital
Locations (1):
- Brigham & Women's Hospital, Boston, Massachusetts, United States